CLINICAL TRIAL: NCT02026336
Title: Inflammatory Asthma Phenotypes Discrimination by an Electronic Nose Breath Analyzer
Brief Title: E-nose and Inflammatory Asthma Phenotypes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Astrid Crespo (Other)
Responsible Party: Sponsor-Investigator, Astrid Crespo, Inflammatory Asthma Phenotypes Discrimination by an Electronic Nose Breath Analyzer, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Organization: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 10/122/1161
Record Dates: First submitted 2013-12-28; First posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Persistent Asthma
Keywords: asthma; inflammation; electronic nose
MeSH Terms: conditions — Asthma; Inflammation | interventions — Electronic Nose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- enose (No Intervention): Electronic nose can discriminate the inflammatory asthma phenotypes, supporting their potential as a non-invasive alternative tool to induced sputum.
  Interventions: Other: electronic nose

INTERVENTIONS:
Other: electronic nose — Exhaled gas to assess e-nose VOC profiles was collected as described. Briefly, patients breathed through a mouthpiece into a 2-way nonrebreathing valve (Hans rudolph 2700, Hans rudolph, Kansas City, Mo) with an inspiratory VOC filter and an expiratory silica reservoir to dry the expired air. Expiratory air was collected in a 10-L "Tedlar bag". Within not more than 10 minutes, the bag was connected to the e-nose device (Cyranose 320®; Smith Detections, Pasadena, CA), provided with a 32 organic polymeric nano-composite sensor array, for 5 minutes and changes in the nano-sensor electrical resistance generated a breath-print VOC profile.
  Other Names: Cyranose 320®; Smith Detections, Pasadena, CA

SUMMARY:
Patients with persistent asthma have different inflammatory phenotypes. The electronic nose is a new technology capable of distinguishing volatile organic compound breath-prints in exhaled breath among different pulmonary diseases.

Question of the study. Is the electronic nose breath-print analysis able to discriminate among different inflammatory asthma phenotypes?

DETAILED DESCRIPTION:
Materials/patients and methods. Fifty-two consecutively enrolled patients with persistent asthma were included in a cross-sectional proof of concept study. Inflammatory asthma phenotypes were recognized by inflammatory cell counts in induced sputum. Breath-prints were analyzed by discriminant analysis on principal component reduction, resulting in cross-validated accuracy values. Receiver Operating Characteristics (ROC) was calculated.

Legal and ethical aspects The study was conducted in accordance with the Declaration of Helsinki principles (18th Word Medical Assembly, 1964) and was approved by the Clinical Research Ethics Committee (approval number: IIBSP/10/122/1161) of our institution. The participants provided their written informed consent to participate in this study and personal identification data were anonymized.

ELIGIBILITY:
Inclusion Criteria:

Adults with persistent asthma, defined as per the Global INitiative for Asthma Management (GINA) criteria, and specifically with positive bronchodilator test, or a daily peak expiratory flow (PEF) variability greater than 20%, or a positive methacholine challenge test documented in case history. Subjects were consecutively enrolled from the outpatient visits of a specialized Asthma Unit located in a tertiary University Hospital.

Exclusion Criteria:

Subjects were excluded if they had a respiratory tract infection or asthma exacerbation within 30 days prior to inclusion or were receiving oral steroids or immunosuppressive treatments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Inflammatory Asthma Phenotypes Discrimination by an Electronic Nose Breath Analyzer | 2 years
  The recognition of volatile organic compound profiles in exhaled air by an electronic nose device can discriminate the inflammatory phenotype of patients with persistent asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Plaza, Principal Investigator — Department of Respiratory Medicine, Hospital de la Santa Creu i Sant Pau. Institut d'Investigació Biomédica Sant Pau (IIB Sant Pau). Universitat Autònoma de Barcelona, Department of Medicine. Barcelona Respiratory Network (BRN). Barcelona, Spain.
Locations (1):
- Vicente Plaza, Barcelona, Spain

REFERENCES:
- [Background] Fens N, Zwinderman AH, van der Schee MP, de Nijs SB, Dijkers E, Roldaan AC, Cheung D, Bel EH, Sterk PJ. Exhaled breath profiling enables discrimination of chronic obstructive pulmonary disease and asthma. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1076-82. doi: 10.1164/rccm.200906-0939OC. Epub 2009 Aug 27. PMID 19713445
- [Background] Dragonieri S, Annema JT, Schot R, van der Schee MP, Spanevello A, Carratu P, Resta O, Rabe KF, Sterk PJ. An electronic nose in the discrimination of patients with non-small cell lung cancer and COPD. Lung Cancer. 2009 May;64(2):166-70. doi: 10.1016/j.lungcan.2008.08.008. Epub 2008 Oct 1. PMID 18834643
- [Background] Petsky HL, Cates CJ, Lasserson TJ, Li AM, Turner C, Kynaston JA, Chang AB. A systematic review and meta-analysis: tailoring asthma treatment on eosinophilic markers (exhaled nitric oxide or sputum eosinophils). Thorax. 2012 Mar;67(3):199-208. doi: 10.1136/thx.2010.135574. Epub 2010 Oct 11. PMID 20937641
- [Background] Executive Committee GEMA 2009. GEMA 2009 (Spanish guideline on the management of asthma). J Investig Allergol Clin Immunol. 2010;20 Suppl 1:1-59. No abstract available. PMID 21413563
- [Background] Montuschi P, Santonico M, Mondino C, Pennazza G, Mantini G, Martinelli E, Capuano R, Ciabattoni G, Paolesse R, Di Natale C, Barnes PJ, D'Amico A. Diagnostic performance of an electronic nose, fractional exhaled nitric oxide, and lung function testing in asthma. Chest. 2010 Apr;137(4):790-6. doi: 10.1378/chest.09-1836. Epub 2010 Jan 15. PMID 20081096
- [Background] Ibrahim B, Basanta M, Cadden P, Singh D, Douce D, Woodcock A, Fowler SJ. Non-invasive phenotyping using exhaled volatile organic compounds in asthma. Thorax. 2011 Sep;66(9):804-9. doi: 10.1136/thx.2010.156695. Epub 2011 Jul 11. PMID 21749985
- [Background] Wenzel SE. Asthma phenotypes: the evolution from clinical to molecular approaches. Nat Med. 2012 May 4;18(5):716-25. doi: 10.1038/nm.2678. PMID 22561835
- [Background] Chung KF, Wenzel SE, Brozek JL, Bush A, Castro M, Sterk PJ, Adcock IM, Bateman ED, Bel EH, Bleecker ER, Boulet LP, Brightling C, Chanez P, Dahlen SE, Djukanovic R, Frey U, Gaga M, Gibson P, Hamid Q, Jajour NN, Mauad T, Sorkness RL, Teague WG. International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma. Eur Respir J. 2014 Feb;43(2):343-73. doi: 10.1183/09031936.00202013. Epub 2013 Dec 12. PMID 24337046
- [Derived] Plaza V, Crespo A, Giner J, Merino JL, Ramos-Barbon D, Mateus EF, Torrego A, Cosio BG, Agusti A, Sibila O. Inflammatory Asthma Phenotype Discrimination Using an Electronic Nose Breath Analyzer. J Investig Allergol Clin Immunol. 2015;25(6):431-7. PMID 26817140
- See also: GINA. Global strategy for asthma management and prevention, global initiative for asthma (GINA) — http://Www.ginasthma.org/.